CLINICAL TRIAL: NCT05504525
Title: Fascia Iliaca Versus Quadratus Lumborum Block for Postoperative Pain Management in Total Hip Replacement: A Comparative Prospective Randomized Study
Brief Title: Fascia Iliaca Versus Quadratus Lumborum Block for Pain Management in Total Hip Replacement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh Refaat, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R118/2021
Record Dates: First submitted 2022-06-04; First posted 2022-08-17 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Opioid Requirements in Patients With Traumatic Fracture Hip
Keywords: opioid requirements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca block for postoperative pain management in hip arthroplasty (Active Comparator)
  Interventions: Procedure: Fascia Iliaca block
- Quadratus lumborum block for postoperative pain management in hip arthroplasty (Active Comparator)
  Interventions: Procedure: Quadratus lumborum block

INTERVENTIONS:
Procedure: Fascia Iliaca block — Ultrasound guided fascia iliaca block done by palpation of anterior superior iliac spine to identify the inguinal crease, then place the ultrasound probe on it to identify the sartorius muscle. Sonographic anatomy will be identified, from superficial to deep, consisting of subcutaneous fat, the internal oblique muscle, the transverse abdominis muscle, the fascia iliaca covering the iliacus muscle and the iliacus muscle itself. The block needle will be advanced in out-of plane to puncture the fascia iliaca. With the needle tip just below the fascia iliaca, 2 ml of a local anesthetic will be injected to confirm the tip location. Once the proper position is confirmed, 40 ml of bupivacaine 0.25% will be injected superficial to the iliacus muscle and deep to the fascia iliaca.
  Arms: Fascia iliaca block for postoperative pain management in hip arthroplasty
Procedure: Quadratus lumborum block — The patients will receive anterior ultrasound guided quadratus lumborum block QLB in the lateral position. The transducer will be first placed in a parasagittal orientation 3-4 cm lateral to the midline and over the sacrum to identify the L5 transverse process. The probe will then rotated into a transverse orientation with slight medial and caudal angulation to obtain a transverse oblique view at L5 transverse process .The ultrasound probe will be tilted , so the lateral end of the probe will be more cranial than the medial side of the probe to avoid the acoustic shadow of the iliac crest. Identify the quadratus lumborum and psoas major and inject the local anesthetic above the QL
  Arms: Quadratus lumborum block for postoperative pain management in hip arthroplasty

SUMMARY:
Postoperative analgesia is essential for early ambulation of patients with hip arthroplasties as well as decreasing hospital stay time. Fascial plane blocks are emerging as a gold standard for postoperative analgesia instead of opioids and NSAIDs, with all there side effects.

The investigators aim to compare postoperative pain levels and opioid analgesic needs of fascia iliaca block versus quadratus lumborum block in patients undergoing primary total hip arthroplasty under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* All patients aging between 40-60 years ASA II, III with no known hypersensitivity for local anesthetics

Exclusion Criteria:

* Patient refusal
* Known allergy to local anesthetics
* Previous femoral artery surgery
* Local infection at the site of injection
* Those on anticoagulation therapy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 24 hours
  The investigators will measure the time to first analgesic request after giving the block

SECONDARY OUTCOMES:
Total rescue analgesic requirements | 24 hours
  Measuring the total rescue analgesic requirement in the postoperative period
Functional recovery | 72 hours
  Will be assessed by duration of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospitals, Cairo, Egypt